CLINICAL TRIAL: NCT01739530
Title: Phase I Study to Evaluate Safety of Repaircell in Healthy Volunteers
Brief Title: Safety of Repaircell in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANT-adip-AL-001
Record Dates: First submitted 2012-11-15; First posted 2012-12-03 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Healthy

ARMS (1):
- Repaircell (Experimental): allogenic differentiated adipocyte
  Interventions: Biological: Repaircell

INTERVENTIONS:
Biological: Repaircell — allogenic differentiated adipocyte

SUMMARY:
Allogenic differentiated adipocytes (ANT-adip-AL) is produced by well-established techniques including cell harvesting from lipoaspirates obtained from healthy donors, expansion of adipose tissue derived stem cells, and differentiation into pure and immature adipocytes. This was an open-label study. Subjects were received subcutaneous injection of ANT-adip-AL and followed for 8 weeks according to the clinical trial protocol.

ELIGIBILITY:
Inclusion Criteria:

* male, 19 years of age or older
* volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening
* informed consent form signed

Exclusion Criteria:

* volunteers who have participated in other clinical studies related cell therapy within 30 days before this clinical trial
* volunteers who received any immune-suppressive drug, corticosteroid or cytotoxic drug within the previous 30 days
* volunteers who have tattoo or scar which disturb assessment of study at injection site
* volunteers who have Creutzfeldt Jacobs disease or related disease or family history
* volunteers who have allergy to bovine-derived materials
* volunteers who have infectious disease such as hepatitis B virus (HBV), hepatitis C virus (HCV)and HIV
* volunteers who have a symptom of septicemia or diagnosis of active Tuberculosis
* volunteers who have a clinically relevant history of abuse of alcohol or drugs
* volunteers who are considered not suitable for the study by investigator
* volunteers who have history of surgery for malignant cancer in the past 5 years
* volunteers who have congenital or acquired immunodeficiency syndrome
* volunteers who have horrible anemia or thrombopenia
* volunteers who have chronic disease such cardiovascular,renal and respirometer disease
* volunteers who were immunosuppressed by disease (ex: chronic heart failure)
* volunteers who were immunodepressed by treatment of medication
* volunteers who is being treated with blood derivatives/who is going to get a blood derivatives
* volunteers who have abnormal rage of CD4/CD8 ratio

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | week 8
  Evaluate the safety at week 8 whether any kind of Adverse event occurs

SECONDARY OUTCOMES:
Immunological response II | week 8
  Infiltration of immune cells by histology based on five basic parameters: (0) No evidence of immune cell infiltration in all area of the tissue, (1) Slight immune cell infiltration visible in partial area of the tissue (barely visible), (2) Obvious immune cell infiltration visible in partial area of the tissue, (3) Slight immune cell infiltration visible in all area of the tissue, and (4) Intense immune cell infiltration visible in all areas of the tissue.
Immunological response I | change from baseline CD4/CD8 ratio at week 8
  CD4 (cluster of differentiation 4)/CD8 (cluster of differentiation 8) ratio

CONTACTS AND LOCATIONS:
Overall Officials: Sa-ik Bang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea